CLINICAL TRIAL: NCT00997269
Title: Benefit of CoQ-10 in Patients on Statins
Acronym: CoQ-10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-0436; AT004204
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Pain; Soreness; Weakness; Fatigue
Keywords: CoQ-10; statin; muscle pain; cardiovascular
MeSH Terms: conditions — Pain; Asthenia; Fatigue; Myalgia | interventions — Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CoQ-10 supplementation (Experimental)
  Interventions: Dietary Supplement: Co-enzyme Q-10
- CoQ-10 placebo supplementation (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Co-enzyme Q-10 — Patients will be supplemented with 300 mg of CoQ-10 1 time daily for one month
  Other Names: ubiquinone
  Arms: CoQ-10 supplementation
Dietary Supplement: Placebo — Patients will be supplemented with CoQ-10 placebo 1 time daily for one month
  Arms: CoQ-10 placebo supplementation

SUMMARY:
This study will investigate whether a supplement called co-enzyme Q10 can help ease or eliminate some of the side effects that result from taking statin medications. These side effects include muscle pain, fatigue or muscle cramping.

DETAILED DESCRIPTION:
Specific Aim 1: to demonstrate that supplementation with coQ10 in patients treated with statins ameliorates symptoms of muscle pain and fatigue and improves energy metabolism and muscle function.

This objective will be achieved in a randomized, placebo-controlled double blind trial by assessing the degree of muscle symptoms and interference of pain with daily activities, aerobic capacity, and muscle function before and after supplementation with either coQ10 or placebo in groups of statin-treated subjects.

Specific Aim 2: to examine changes at a molecular/cellular level that are associated with improved pain and muscle function in statin-treated subjects supplemented with coQ10.

This aim will be addressed by analyzing muscle biopsies taken from statin-treated patients before and after supplementation with coQ10 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women 21 years and older taking statin medications for hyperlipidemia under the current National Cholesterol Education Program guidelines (NCEP III) and complaining of myopathic symptoms.

Exclusion Criteria:

1. diagnosis of cancer;
2. acute illness of any sort;
3. hemoglobin less than 12,
4. creatinine greater than 1.5 mg/dl;
5. liver dysfunction as evidenced by elevations in transaminases 3-fold higher than upper limit of normal;
6. use of certain medications or nutritional supplements within the past month;
7. untreated hypertension (diastolic BP> 100 mm HG);
8. diagnosis of diabetes mellitus (fasting blood glucose > 126 mg/dl);
9. untreated hypothyroidism;
10. overt congestive heart failure (by physical exam);
11. active inflammatory diseases such as rheumatoid arthritis, lupus, etc.,
12. bleeding disorders;
13. history of adverse reactions besides myopathy associated with the use of statins;
14. any previous adverse reaction to coQ10 or to multivitamin supplements containing coQ10;
15. plasma CPK levels > 3 times the upper normal limit; OR
16. congenital myopathies and/or neuromuscular degenerative diseases.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain scores should be reduced | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Caso, MD, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University GCRC, Stony Brook, New York, United States